CLINICAL TRIAL: NCT01443533
Title: A Randomized Controlled Trial of a Brief Educational Script on Postpartum Contraceptive Uptake
Brief Title: Study of Birth Control Use After Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WakeMed Health and Hospitals (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Jennifer H. Tang, Principal Investigator, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WakeMed 864
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Contraception
Keywords: Contraception; Contraception behavior; Postnatal care; Health education; Randomized controlled trial
MeSH Terms: conditions — Contraception Behavior; Health Education

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LARC script (Experimental): Received routine postpartum counseling and LARC script.
  Interventions: Behavioral: LARC Script
- No LARC script (No Intervention): Received only routine postpartum counseling

INTERVENTIONS:
Behavioral: LARC Script — The LARC Script is a one-minute educational script that describes long-acting reversible contraceptive methods.
  Arms: LARC script

SUMMARY:
This study is a randomized controlled trial that will evaluate the impact of a brief educational script on the method of birth control that women receive at their 6-week postpartum visit. The one-minute script ("LARC script") is given to women in the hospital during their postpartum admission. It informs patients about long-acting reversible contraceptive (LARC) methods, specifically the contraceptive implant and the intrauterine device. The investigators hypothesize that women who are randomized to receive the LARC script will be more likely to report that they are using a LARC method, when queried immediately after their six-week postpartum visit.

ELIGIBILITY:
Inclusion Criteria:

* Women who are admitted to the postpartum unit at WakeMed Hospital
* Delivery of a live infant >24 weeks gestational age
* Age 14-45 years
* Ability to speak either English or Spanish fluently
* Willing to be contacted by phone until at least 8 weeks after delivery

Exclusion Criteria:

* History of a tubal ligation or hysterectomy
* Partner has already had a vasectomy
* History of fertility treatment to conceive this pregnancy
* Previous randomization into the study

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 800 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Self-reported use of LARC method | After six-week postpartum visit

SECONDARY OUTCOMES:
Self-reported interest in use of a LARC method | After six-week postpartum visit
Self-reported use of any contraceptive method | After six-week postpartum visit
Self-reported reasons for not using the contraceptive method of choice | After six-week postpartum visit

CONTACTS AND LOCATIONS:
Locations (1):
- WakeMed Hospital, Raleigh, North Carolina, United States

REFERENCES:
- [Background] Secura GM, Allsworth JE, Madden T, Mullersman JL, Peipert JF. The Contraceptive CHOICE Project: reducing barriers to long-acting reversible contraception. Am J Obstet Gynecol. 2010 Aug;203(2):115.e1-7. doi: 10.1016/j.ajog.2010.04.017. Epub 2010 Jun 11. PMID 20541171
- [Background] Lopez LM, Hiller JE, Grimes DA. Postpartum education for contraception: a systematic review. Obstet Gynecol Surv. 2010 May;65(5):325-31. doi: 10.1097/OGX.0b013e3181e57127. PMID 20591202
- [Background] Stanwood NL, Bradley KA. Young pregnant women's knowledge of modern intrauterine devices. Obstet Gynecol. 2006 Dec;108(6):1417-22. doi: 10.1097/01.AOG.0000245447.56585.a0. PMID 17138775
- [Background] Conde-Agudelo A, Rosas-Bermudez A, Kafury-Goeta AC. Birth spacing and risk of adverse perinatal outcomes: a meta-analysis. JAMA. 2006 Apr 19;295(15):1809-23. doi: 10.1001/jama.295.15.1809. PMID 16622143
- [Derived] Zerden ML, Tang JH, Stuart GS, Norton DR, Verbiest SB, Brody S. Barriers to Receiving Long-acting Reversible Contraception in the Postpartum Period. Womens Health Issues. 2015 Nov-Dec;25(6):616-21. doi: 10.1016/j.whi.2015.06.004. Epub 2015 Jul 23. PMID 26212318